CLINICAL TRIAL: NCT03469362
Title: Randomized Clinical Trial of Intracorporeal vs Extracorporeal Urinary Diversion After Robot Assisted Radical Cystectomy
Brief Title: Intracorporeal vs Extracorporeal Urinary Diversion After Robot Assisted Radical Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Mark L. Gonzalgo, MD, PhD, Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20170004
Record Dates: First submitted 2018-03-06; First posted 2018-03-19 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-11

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Extracorporeal Urinary Diversion (ECD) (Experimental): Participants will be randomized to receiving ECD after scheduled Robotic Assisted Radical Cystectomy (RARC).
  Interventions: Procedure: Extracorporeal Urinary Diversion
- Intracorporal Urinary Diversion (ICD) (Experimental): Participants will be randomized to receiving ICD after scheduled Robotic Assisted Radical Cystectomy (RARC).
  Interventions: Procedure: Intracorporal Urinary Diversion

INTERVENTIONS:
Procedure: Extracorporeal Urinary Diversion — Extra-corporeal urinary diversion, provided as part of standard of care, will have the ureters sutured into the ileal conduit by hand.
  Other Names: ECD
  Arms: Extracorporeal Urinary Diversion (ECD)
Procedure: Intracorporal Urinary Diversion — Intracorporal Urinary Diversion, provided as part of standard of care, will have the ureters sutured into the ileal conduit using the Da Vinci robot.
  Other Names: ICD
  Arms: Intracorporal Urinary Diversion (ICD)

SUMMARY:
Intracorporeal urinary diversion (ICD) provides superior postoperative outcomes compared to extracorporeal urinary diversion (ECD). The investigators' hypothesis that ICD may provide clinical benefit is based on principles of less bowel and ureteral handling, superior operating room workflow, less exposure to the external environment, and optimal visualization with ICD while utilizing a smaller incision compared to ECD. ICD should have less bowel-related complications, lower pain scores allowing patients to be discharged from the hospital sooner and regain functional independence more quickly.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven urothelial cancer being considered for RARC.
* Clinical stage T1-T4, N0-1, M0 or refractory carcinoma in situ.
* Subject must be already scheduled to have a RARC at the discretion of the surgeon and with the patient's agreement.

Exclusion Criteria:

* Inability to give informed consent
* Prior major abdominal and pelvic open surgical procedures that would preclude a safe robotic approach, as determined by the treating surgeon.
* At the discretion of the treating surgeon, any pre-existing condition such as severe chronic obstructive pulmonary disease that precludes a safe initiation or maintenance of pneumoperitoneum over a prolonged period of time and during surgery.
* Age <18 or >99 years.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
90-day Major Post-Operative Complication Rate | 90 days
  Major complication rate at 90-days from RARC + urinary diversion using the modified Clavien-Dindo grading system. Major complication is defined as Clavien-Dindo Grade ≥ 3.

SECONDARY OUTCOMES:
90-day Any Post-Operative Complication Rate | 90 days
  Any complication rates at 90-days from RARC + urinary diversion, using the modified Clavien-Dindo grading system as low grade (1-2) or high grade (3-5).
Length of Hospital Stay in ECD vs ICD Study Participants | About 2 weeks
  Length of hospital stay for study participants undergoing ECD versus ICD urinary diversion post-RARC, as recorded at hospital discharge.
90-day Readmission Rate | 90 days
  Rate of readmission to hospital at 90 days post-RARC followed by ECD or ICD urinary diversion.
Rate of Return to the Operating room within 90 days | Up to 90 days
  Rate of return to the operating room within 90 days after RARC followed by ICD or ECD Urinary Diversion.
Mortality Rate at 90 days | 90 days
  Rate of mortality (death) at 90 days in study participants
Rate of Bowel-Specific Complications | Up to 36 months
  Rate of bowel-specific complications in study participants (including incidence of mechanical bowel obstruction, anastomotic leaks, and surgical site infections) and post operative pain. Bowel-specific complications will be assessed using the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 4.
Functional Independence Recovery as measured by the ADL Questionnaire | Up to 36 months
  Rate of functional independence recovery as measured by patient-reported scores on the Activities of Daily Living (ADL) questionnaire. For the ADL, the total score ranges from 0 to 6, with the higher scores indicating functional improvement and lower scores indicating functional deterioration.
Functional Independence Recovery as measured by the IADL Questionnaire | Up to 36 months
  Rate of functional independence recovery as measured by an aggregate of patient-reported scores on the Instrumental Activities of Daily Living (IADL) questionnaire. For the IADL, the total score ranges from 0 to 8, with higher scores indicating functional functional improvement and lower scores indicating functional deterioration.
Functional Independence Recovery as measured by the Hand Grip Strength Test. | Up to 36 months
  The Hand Grip Strength Test measures the amount of static force that a participant's hand can squeeze around a dynamometer. The test is measured in kilograms.
Functional Independence Recovery as measured by the Timed Up and Go (TUG) Walking Test | Up to 36 months
  The TUG test times participants as they rise from a standard chair, walk 3 meters, turn, walk back and sit again. The test is measured in seconds.
Health-Related Quality of Life (HRQoL) as assessed by SF-8 Health Survey | Up to 36 months
  HRQoL measured by patient scores on the Short Form 8 (SF-8) Health Survey. The SF-8 is a questionnaire consisting of 8-items and two component summary scores: Physical component summary (PCS) and mental component summary (MCS). They are scored by weighting each score to a norm-based scoring model. The total scores will be reported as a percentile with higher score indicating better health-related quality of life.
HRQoL as assessed by the FACT-VCI Questionnaire | Up to 36 months
  HRQoL measured by patient scores on the Functional Assessment of Cancer Therapy-Vanderbilt Cystectomy Index (FACT-VCI) questionnaire. The FACT-VCI is a condition-specific instrument for patients undergoing radical cystectomy (RC) and urinary diversion (UD) for bladder cancer. The questionnaire consists of 44 items scored on a range from 0 ("Not at all") to 4 ("Very Much"), resulting in an ordinal Likert scale, with higher scores indicating a better HRQoL. The FACT-VCI measures quality of life across five domains: Physical wellbeing, social/family wellbeing, emotional wellbeing, functional wellbeing and an additional concerns subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Gonzalgo, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No